CLINICAL TRIAL: NCT06392997
Title: Evaluation of Salivary RNA in Subjects Scheduled for Surgery for a Gynecologic Pathology
Acronym: GynRNA
Status: Recruiting | Type: Observational
Sponsor: ZIWIG (Industry)
Collaborators: Monitoring Force Group (Industry)
Responsible Party: Sponsor
Other Study IDs: ZWG-24-01
Record Dates: First submitted 2024-04-09; First posted 2024-05-01 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Gynecologic Disease; Gynecologic Cancer; Endometriosis; Ovarian Cancer; Cyst Ovary; Fibroid; Cervical Cancer; Uterine Cancer
MeSH Terms: conditions — Genital Diseases, Female; Endometriosis; Ovarian Neoplasms; Ovarian Cysts; Leiomyoma; Uterine Cervical Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salivary samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Symptomatic group: Clinically symptomatic females with one or more of the following gynecological pathology:
  * Endometriosis,
  * Adenomyosis,
  * Ovarian cysts,
  * Fibroids,
  * Ovarian cancer,
  * Cervical cancer
  * Uterine cancer.
  Interventions: Diagnostic Test: Saliva sample
- Asymptomatic group: Asymptomatic females with:
  * Cervical dysplasia or cancer
  * A normal pap-smear (control)
  Interventions: Diagnostic Test: Saliva sample

INTERVENTIONS:
Diagnostic Test: Saliva sample — Saliva sample

SUMMARY:
GynRAN is an international, multicentre, transversal, diagnostic and non-interventional study carried out in gynecology-obstetrics/gynecological oncology departments that aims to identify a diagnostic signature for gynecological pathologies by analyzing of coding and non-coding RNA contained in patients saliva.

The study population consists of patients with clinically symptomatic females with one or more of the gynecological pathologies (endometriosis, adenomyosis, ovarian cysts, fibroids, ovarian/cervical/uterine cancer) and asymptomatic females.

The patients concerned by the study will be managed without modification of the care pathway, nor modification of the therapeutic indications, nor modification of the diagnostic or follow-up examinations necessary according to the context, which are carried out according to the local recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Subject of legal age (according to local legislation) and at least 18 years old
2. Subject (and if applicable her legal representative) having dated and signed the informed consent form
3. Subject with a medical insurance policy
4. Subject presenting to the department:

   1. With Symptoms (bleeding and/or pain and/or clinically observed symptom) of one or more of the following pathologies (suspected undergoing diagnostic surgery/biopsy or diagnosed and before any curative treatment of the pathology):

      * Endometriosis
      * Adenomyosis,
      * Ovarian cysts,
      * Fibroids,
      * Ovarian cancer,
      * Cervical cancer,
      * Uterine cancer.
   2. Asymptomatic with pap smear positive for cervical dysplasia or cervical cancer and before any curative treatment.
   3. Asymptomatic undergoing a pap smear for cervical cancer screening in a gynecological follow-up context.

Exclusion Criteria:

1. Recent (<1 month) or ongoing bacterial or viral infection
2. Known active oral or digestive mycosis
3. Evolving oral pathology, symptomatic or obvious
4. Known pregnancy
5. Known current non-gynecological pelvic pathology
6. Subject with a diagnosed breast cancer or cancer other than gynecological with the exception of basal cell carcinoma
7. Subject with a history of treated cancer within the last 5 years with the exception of basal cell carcinoma
8. Subject who has already received chemotherapy or radiotherapy or undergone complete or partial excision of the gynecological pathology of inclusion criterion
9. Subject with significant difficulties reading or writing her language
10. Subject unable to comply with study and/or follow-up procedures
11. Participation in an interventional study with investigational drug or in the exclusion period of an interventional study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study populations is constituted of s:
  1. Clinically symptomatic females with one or more of the following gynecological pathology:
     * Endometriosis,
     * Adenomyosis,
     * Ovarian cysts,
     * Fibroids,
     * Ovarian cancer,
     * Cervical cancer
     * Uterine cancer.
  2. Asymptomatic females with:
     * cervical dysplasia or cancer
     * a normal pap-smear (control)
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the Receiver Operating Curve (ROC) | Through the end of study inclusions, an average of 1 year
  Identify a diagnostic signature for each pathology (Endometriosis / Adenomyosis / Ovarian cysts / Fibroids / Cervical Displasia / Ovarian cancer / Cervical cancer /Uterine cancer) by analyzing of coding and non-coding RNA contained in the saliva.

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU d'Angers, Angers
  - Clinique Tivoli Ducos - IFEMENDO, Bordeaux
  - Institut Bergonié, Bordeaux
  - CHU Caen, Caen
  - CGFL, Dijon
  - CHU Lyon Sud, Lyon
  - American Hospital of Paris, Neuilly-sur-Seine
  - CHU de Rennes Site Hôpital Sud, Rennes
  - Clinique La sagesse, Rennes
  - CHU Rouen, Rouen
  - Clinique Pasteur, Toulouse
  - CHU Bretonneau-Tours, Tours
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No